CLINICAL TRIAL: NCT00154076
Title: A Multicenter Comparative Trial of Zonisamide and Topiramate as Initial Monotherapy in Untreated Epilepsies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Jihee Mun, Eisai Korea Inc.
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2090-S082-403
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide; Topiramate

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Zonisamide
- 2 (Active Comparator)
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Zonisamide — Initial dose is 100mg/day, increase after 2 weeks to 200mg/day. The maximum dose is 600mg/day.
  Other Names: Zonegran
  Arms: 1
Drug: Topiramate — Initial dose is 25mg/day, increase every 1 week to 100mg/day. The maximum dose is 400mg/day.
  Arms: 2

SUMMARY:
To assess the efficacy and safety of Zonisamide and Topiramate as Initial Monotherapy in Untreated Epilepsies

ELIGIBILITY:
Inclusion criteria:

1. Patients over 13 years old (complete the elementary school course).
2. Patients had at least two seizures in the past and at least one seizure for the last 3 months before screening.
3. Patients had no antiepileptic drugs for the last 4 months.
4. Women of childbearing age who agree to contraception during participating this clinical trial.

Exclusion criteria:

1. Pregnancy
2. Patients who have progressive neurologic disease
3. Allergy to sulfonamides
4. Use of acetazolamide within a year
5. Hemolytic anemia
6. Patients who have abnormal liver function (GOT or GPT) values more than twice the normal values.
7. Patients who have abnormal renal function (BUN or Creatinine) values more than three times the normal values.
8. Patients who have history of drug or alcohol abuse.
9. Glucose-6-phosphate dehydrogenase deficiency.
10. Patients who were detected with renal stones on KUB (Kidney-Ureter-Bladder) test.
11. Patients who have progressive internal or surgical disease.
12. Patients who have progressive psychiatric disease.
13. Patients who have mental retardation (IQ 70 and less).
14. Patients taking Vit C.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | 2, 4, 8, 12, 16, 20, 24 weeks

SECONDARY OUTCOMES:
Cognitive function | 0, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jihee Mun, Study Director — Eisai Korea Inc.
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea